CLINICAL TRIAL: NCT05358262
Title: Using Highly Heated Humidification to Minimize Aerodigestive Tract Complications of Autologous Stem Cell Transplant
Brief Title: High Heated Humidity in Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0017
Record Dates: First submitted 2022-04-19; First posted 2022-05-03 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Autologous Stem Cell Transplant
Keywords: Mucositis
MeSH Terms: conditions — Mucositis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention using the Airvo device (Experimental): Patients randomized to this group will receive the standard of care as well as wear the Airvo (equipment to provide high heated humidity) starting on Day 0 of their transplant for a minimum of 4 hours a day (to be worn in one continuous block of time). The humidity is delivered by nasal cannula that goes into your nose, similar to wearing oxygen. The equipment stands on a pole and plugs into a power outlet. Patients may take off the equipment for short periods of time. Eg to go to the bathroom.
  Interventions: Device: Airvo
- Standard of Care (Active Comparator): Patients randomized into this group will receive the usual standard of care for mucositis.
  The standard of care for mucositis at the Cross Cancer institute involves supportive therapies including oral hydration (water or wet sponges) or medicated mouthwashes.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Airvo — Fisher & Paykel's AIRVO 2 is a humidifier with integrated flow generator that delivers high flow warmed and humidified respiratory gases to spontaneously breathing patients through a variety of interfaces including nasal cannula. Flow can be delivered from 2 to 60 LPM
  Arms: Intervention using the Airvo device
Other: Standard of Care — The standard of care for mucositis at the Cross Cancer institute involves supportive therapies including oral hydration (water or wet sponges) or medicated mouthwashes.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to find out what effects of high heated humidity has on you and your mucositis.

DETAILED DESCRIPTION:
This is a open label, case-control randomized, phase II clinical trial comparing the use of High Heated Humidity (H3) delivered using the Airvo 2 device to standard of care in Hematologic cancer recipients of autologous stem cell transplant (including Hodgkin lymphoma, non-Hodgkin lymphoma, and multiple myeloma).

Mucositis and aerodigestive tract complications are common across most types of cytotoxic chemotherapies. These complications are both more frequent and severe in recipients of high dose chemotherapy (HDT) and autologous stem cell transplant (ASCT). By extending the use of H3 to include the HDT/ASCT population, there is the possibility to decrease or minimize the complications associated with the current standard treatment process. Shorter, less complicated hospital stays could results for those whose course would otherwise end up being longer due to complications/set- backs. The length of time to use the device per day is a minimum of 4 hours/day up to approximately 14 days while being an inpatient. Treatment beyond 14 days is exceptional and will be done only in those individuals who continue to have mucositis beyond 14 days. In this case, patients may receive treatment up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 18 years of age
2. Have given written consent prior to any study-specific procedures or have had an acceptable individual capable of giving consent on the patient's behalf.
3. Have one of non-Hodgkin lymphoma, Hodgkin lymphoma, or multiple myeloma and found to require high-dose, melphalan-based chemotherapy and autologous stem cell transplant (ASCT) as part of standard of care treatment (includes patients receiving ASCT also requiring oxygen).
4. Performance status of ECOG 0-2
5. Are reliable and willing to make themselves available for the duration of the study, and are willing to follow study procedures.

Exclusion Criteria:

1. Nasal blockage such as nasal polyps, deviated septum or nasal packing would either not allow the proper flow of heated humidity into the nares or it would be too uncomfortable to tolerate during the intervention.
2. Those with influenza like illness. The intervention is not in itself, an aerosol generating medical device. However, if influenza positive, there could be airborne spread of the virus impacting both staff and other patients.
3. Tracheostomy Tube Patients would require a different type of equipment attachment which is not included in this study. Tracheostomy tubes by-pass the upper airway and therefore the intervention cannot be used for the purpose of assessing mucositis. This intervention is used regularly on tracheostomy patients with good success however in this case, the upper airway is by-passed and therefore there would be no impact on mucositis.
4. Patients with significant co-morbidities that would prevent compliance of equipment use as determined by the treating physician.
5. Patients who have Obstructive Sleep Apnea who use a CPAP machine at night. This population would not be able to use the intervention concurrently with the CPAP device as both utilize the nares.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mucositis severity symptoms | During treatment (up to 30 days)
  Mucositis is defined as inflammation of the oral and aerodigestive tract mucosa. Patient subjective measure, such as patient reported discomfort or sensation of inability to clear secretion will be observed using the Oral Mucositis Quality of Life Questionnaire.
Mucositis severity assessment | During treatment (up to 30 days)
  Mucositis is defined as inflammation of the oral and aerodigestive tract mucosa. Patient objective measures, such as increased reddening of the mucosa to ulcerations will be observed using the Oral Assessment Guide.

SECONDARY OUTCOMES:
Febrile Neutropenia | During treatment (up to 30 days)
  To minimize febrile neutropenia which is low neutrophil count with fever.
Nosocomial infections | During treatment (up to 30 days)
  To minimize infections during stay in hospital.
Length of stay to be changed in hospital | During treatment (up to 30 days)
  To minimize hospital stay when infection decreased
Dietary pattern/intake | During treatment (up to 30 days)
  Because of the direct effect of mucositis on the ability to eat and drink, dietary intake/pattern and weight is likely to be impacted.The 31-point Oral Mucositis Quality of Life (OMQoL) scale is to be used while patients are receiving H3 treatment to subjectively assess patient's dietary quality of life.
Patient weight | The comparison will be weight at admission vs weight at discharge (Day 14 or Day 30)
  Because of the direct effect of mucositis on the ability to eat and drink, dietary intake/pattern and weight is likely to be impacted.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Lem, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No